CLINICAL TRIAL: NCT06025617
Title: Comprehensive Evaluation of a New Diagnostic Clinic for Functional Disorders - the DISTRESS Trial
Brief Title: DISTRESS Trial Functional Disorders - the DISTRESS Trial
Acronym: DISTRESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regionshospitalet Silkeborg (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Michael Moesmann Madsen, Clinical assistant and Medical Doctor, Regionshospitalet Silkeborg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 147304
Record Dates: First submitted 2023-08-07; First posted 2023-09-06 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Bodily Distress Syndrome; Functional Somatic Disorder
Keywords: Fibromyalgia; Irritable Bowel Syndrome; Chronic Fatigue Syndrome; Somatoform Disorders
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic; Somatoform Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Outcome data is blinded to the investigator during data analysis as to intervention vs. comparison arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Patients referred by their GP under suspicion of suffering from FSD are randomized to the intervention arm.
  Interventions: Other: Diagnostic evaluation at the Diagnostic Clinic for Functional Disorders
- Control arm (Active Comparator): Patients referred by their GP under suspicion of suffering from FSD are randomized to "Diagnostic as usual" in the control arm.
  Interventions: Other: Diagnostic as usual

INTERVENTIONS:
Other: Diagnostic evaluation at the Diagnostic Clinic for Functional Disorders — The intervention consists of being examined at the Diagnostic Clinic for Functional Disorders. If an FSD diagnosis is established, the patient receives feed-back of on the FSD diagnosis and patient education about the condition. Subsequently, the clinic provides guidance to the GP regarding recommended management and treatment options tailored to each individual patient.
  Arms: Intervention arm
Other: Diagnostic as usual — "Diagnostic as usual" consists in being referred to be examined at another existing specialist clinic in the secondary sector, as specified by the patient's GP.
  Arms: Control arm

SUMMARY:
A Diagnostic Clinic for Functional Somatic Disorders (FSD) has been set up at the outpatient diagnostic center at Regionshospitalet Silkeborg. The objective of the clinic is to support General Practitioners (GPs) by offering early stage diagnostic evaluation of whether a patient has an FSD or the symptoms were caused by another physical illness or mental disorder.

As a novelty in this project, Internal Medicine consultants examine the patients for FSD, after having received training in diagnosing FSD by FSD experts. By performing diagnostic evaluation for physical diseases and FSD simultaneously, the investigators believe that the new clinic shall be able to accelerate the establishment of a final diagnosis for these patients who would otherwise likely undergo a protracted diagnostic course involving sequential evaluations at various specialty clinics.

The DISTRESS trial is a pragmatic randomized clinical trial which aims to evaluate the Diagnostic Clinic for FSD in terms of clinical cost-effectiveness outcomes.

DETAILED DESCRIPTION:
Functional Somatic Disorders (FSD) are conditions where patients present with characteristic patterns of physical symptoms, accompanied by impairment or disability. FSD is a clinical diagnosis for which no clinical or paraclinical tests at present have been found useable for establishing the diagnosis. The disorders range from mild and transient to severe, chronic and disabling, and are common in all medical settings, both in primary and secondary care. FSD is costly for society due to high health care use, and the reduction of patients' labor market participation. Arguably, insufficient diagnostic availability is part of the reason some patients develop more severe, chronic and disabling FSD. The Diagnostic Clinic for FSD was set up at Regionshospitalet to alleviate this diagnostic need in the secondary care setting.

The DISTRESS trial is a pragmatic randomized clinical trial. After referral by their GP, patients are randomized 1:1 into two study arms: Intervention and Control. The referring GP must specify which diagnostic evaluations he/she requests both in the intervention and in the control group.

Intervention arm: Patients in this arm shall be examined by an internal medicine specialist trained in FSD diagnostic evaluation at The Diagnostic Clinic for FSD. After parallel evaluation for FSD and other physical conditions, patients are given their diagnosis, along with patient education in what FSD is, as well as a letter to their GP regarding recommended management and treatment options.

Control arm: The comparison group in the randomized clinical trial will receive diagnostic as usual at the Diagnostic center or elsewhere in the secondary sector in The Central Denmark Region.

In this clinical trial, the investigators aim to evaluate the effectiveness in terms of health-related utility improvement for the patients as well as the healthcare and societal costs and cost-effectiveness of the clinic, compared to diagnostic as usual.

ELIGIBILITY:
Study population:

Participants were drawn from the population of the Central Denmark Region. To be considered for inclusion, patients had to be referred by their GP.

Inclusion Criteria:

* Being referred to the clinic by their GP due to symptoms consistent with a possible diagnosis of moderate or severe FSD.
* Symptoms having been present for at least 6 months and no more than 3 years.
* Having undergone at least 2 diagnostic evaluations (e.g. imaging studies or specialist evaluations) at physical specialty clinics or hospitals in the past year.
* Age 18-60.
* Being of ethnic western cultural upbringing.
* Understands and speaks Danish fluently.

Exclusion Criteria:

* Having another severe chronic disease which explains the reduced level of functioning.
* Having been previously referred to or evaluated for FSD at this or another clinic specializing in functional disorders.
* Previous diagnosis of FSD.
* Alcohol or other substance-dependency or -abuse.
* Emergent psychiatric illness or emergent elevated risk of harm to self or others requiring psychiatric evaluation for possible need of acute or sub-acute psychiatric hospitalization.
* Current or prior diagnosis of psychosis (ICD10 F2x diagnosis), bipolar affective disorder (ICD10 F31.x diagnosis) or depression with psychotic symptoms (ICD10 F32.3 or F33.3 diagnosis).
* Currently pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Healthcare services utilization (i.e. direct costs) | 12 months prior to randomization and 12 months' follow-up
  Comparison of healthcare services utilization (of secondary and tertiary sector care) by the intervention group, compared to the control group. Data shall be drawn from Danish national and regional healthcare service registers.
Cost-effectiveness analysis (CEA) (direct and indirect costs) | 12 months prior to randomization and 12 months' follow-up
  Cost-effectiveness analysis (CEA), comparing the intervention and the control group from both a healthcare (direct costs) and a societal perspective (indirect costs) combining data on incremental costs and incremental effects; adjusted for differences in mean utility score and mean costs at baseline (1 year prior to randomization).

SECONDARY OUTCOMES:
Public expenses associated with occupational status and social benefits (i.e. indirect costs) | 12 months prior to randomization and 12 months' follow-up
  Comparison of expenses associated with occupational status and social benefits of the intervention group, compared to the control group. Data shall be drawn from the Danish Register-based Evaluation of Marginalisation (DREAM) database.
Effectiveness: Health-related quality of life (via the the Short Form 36 Total Score) | Baseline, 3- and 12-months' follow-up
  Difference between the intervention group and the control group in health-related quality of life, measured by the Total Score of the Short Form 36 (SF-36). The SF-36 is summarized in a score on a scale from 0-100 where 100 is the best possible health-related quality of life.
Effectiveness: Perceived physical health | Baseline, 3- and 12-months' follow-up
  Difference between the intervention group and the control group in perceived physical health, measured by an aggregate score of the 'physical functioning', 'bodily pain' and 'vitality' subscales of the Short Form-36. This aggregate score has a minimum of 15 and a maximum of 65 and a higher score indicates better physical health. This outcome encompasses physical domains which have been previously found to be affected in functional somatic disorders.
Effectiveness (via Patient-reported Clinical Global Improvement) | At 3- and 12-months' follow-up
  Patients evaluate their overall health as "much worse", " somewhat worse ", "about the same", "somewhat better" or "much better" compared to 1 year prior, at 3 and 12 months after randomization. Specifically, we shall compare the share of patients in the intervention group vs. the control group who evaluate their overall health as "somewhat better" or "much better".

OTHER OUTCOMES:
Symptom level comparison | At 3- and 12 months follow-up
  Comparison of the intervention group and the control group regarding the number and severity of symptoms via the Bodily Distress Syndrome 25 (BDS-25) symptom checklist. This checklist asks 'have you been bothered by', followed by a list of 25 symptoms comprising the four symptom clusters of Bodily Distress Syndrome (BDS). The checklist measures symptoms on a 5-point rating scale from 0 ('not at all bothersome') to 4 ('a lot bothersome'). The sum score is calculated by adding the single item scores from the 25 items (ranging from 0 to 100, where a higher score implies greater bother from symptoms).
Health anxiety | At 3- and 12 months follow-up
  Comparison of the intervention group and the control group regarding health anxiety using Whiteley-6-R index. The Whiteley indices measure health anxiety. The Whiteley-6-R, which excludes two items on somatic symptoms while adding one item on obsessive rumination has been found to have better psychometric properties. The Whiteley-6-R has a total score range of 0-24, where a higher score indicates a higher level of health anxiety.
Overall physical health | At 3- and 12 months follow-up
  Overall health is assessed with a single item from the 36-item Short-Form Health Survey (SF-36), estimating self-perceived health on a 5-point rating scale from 'excellent' to 'poor'. Higher score on this item indicates poorer health.

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Madsen, MD MPH MSc, Principal Investigator — Regionshospitalet Silkeborg; Lise K Gormsen, MD PhD, Study Chair — Funktionelle Lidelser, Aarhus Universitetshospital; Christian Trolle, MD PhD, Study Director — Regionshospitalet Silkeborg; Per Fink, MD Dr. Med PhD, Study Director — Funktionelle Lidelser, Aarhus Universitetshospital
Locations (1):
- Regionshospitalet Silkeborg, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madsen MM, Trolle C, Fynne LV, Colombo M, Pedersen RL, Sorensen VN, Christensen SR, Fink P, Gormsen LK. Early identification of functional somatic disorders in an internal medicine diagnostic clinic: The DISTRESS trial. Contemp Clin Trials. 2025 Nov;158:108082. doi: 10.1016/j.cct.2025.108082. Epub 2025 Sep 17. PMID 40972891